CLINICAL TRIAL: NCT02330354
Title: Our Year of Healthy Living: A Social Marketing Intervention for Child Care & Home
Brief Title: Our Year of Healthy Living (Formative Research & Intervention)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 13-2379; R01HL120969 (NIH)
Record Dates: First submitted 2014-12-23; First posted 2015-01-01 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: preschool; behavior change; social marketing; child care providers; nutrition; child care centers; physical activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Centers in this group will participate in the Healthy Me, Healthy We program.
  Interventions: Behavioral: Healthy Me, Healthy We
- Control Group (Other): Centers in this group will participate in the Healthy Me, Healthy We program after follow-up measures are collected.
  Interventions: Behavioral: Healthy Me, Healthy We

INTERVENTIONS:
Behavioral: Healthy Me, Healthy We — The intervention - Healthy Me, Healthy We - is a 7-month social marketing campaign designed to improve preschool children's (3-4 years) diet and physical activity behaviors.

SUMMARY:
The purpose of this study is to evaluate the effect of a 7-month social marketing program - Healthy Me, Healthy We (previously called Our Year of Healthy Living) - in improving preschool children's (3-4 years) diet and physical activity behavior. Healthy Me, Healthy We will use social marketing approaches in the child care center to promote the use of healthy diet and physical activity behaviors by children, as well as their teachers and parents. The program will use visual cues, educational materials, activities, and a song to deliver targeted healthy behavior messages that connect the teacher, child, and parents. Centers will implement the Our Year of Healthy Living program in their classrooms over the course of a school year (October-April). Prior to initiation and after completion of the program, researchers will collect information about diet, physical activity, child body mass index (BMI), and center and home environment information from participants. From the beginning of the program to the end, children enrolled in the program will have 1) a greater increase in physical activity and decrease in sedentary time, 2) improved diet, and 3) smaller increase in body mass index compared to children in centers that do not complete the program. Additionally, from the beginning of the program to the end, homes and centers that participate in the program will have greater improvements in scores on the home and center environment assessments compared to centers and homes that do not participate.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of the 7-month social marketing intervention - Healthy Me, Healthy We (previously called Our Year of Healthy Living) - in improving preschool children's (3-4 years) diet and physical activity behaviors. The study will use a two-arm, cluster randomized controlled design and a sample of 90 child care centers and 810 children (9 parent-child dyads/center).

For this study, the investigators will recruit 90 child care centers from a mix of urban/suburban and rural areas. Potential child care centers in these counties will be identified using an online database of licensed child care facilities maintained by the North Carolina (NC) Division of Child Development and Early Education. State and local community partners will be engaged to help inform centers in targeted counties about the study. Direct recruitment of centers will employ a variety of strategies (e.g., mail, email, telephone, in-person contacts). Once a center expresses interest, the investigators will work with the center director to recruit nine parent-child dyads and five teachers from the 3- and 4-year old classrooms.

Outcome Measures:

A series of measurements will be collected on participating children, parents, and child care providers at two time points - baseline and follow-up. Primary outcomes measures will assess child physical activity and diet quality. Secondary outcomes measures will assess child weight, center and home environment. These measures will be collected in large part during two-day on-site visits to the child care center, and supplemented with self-administered surveys. Center visits will be conducted by data collectors who have undergone extensive training and certification on all measurement procedures and are blinded to study-arm assignment. Identical data collection protocols will be used at baseline and follow-up.

Children's physical activity will be measured using accelerometers. A data collector will fit each participating child with an accelerometer on a belt during the morning of the first day of the center visit. The child will wear the accelerometer for seven full days - both at child care and at home. Once data are downloaded, age-appropriate cut-points will be applied in order to calculate daily minutes of non-sedentary physical activity.

Children's dietary intakes will be measured using a combination of direct observation and food diaries. The Dietary Observation for Child Care (DOCC), (Ward et al. 2008) will be used to assess foods consumed by children while at child care. Each data collector can assess up to three children at a time; therefore, a team of three data collectors will be assigned to each center to allow observation of the nine participating children. They will observe intakes on two consecutive weekdays, recording all foods and beverages consumed by the children during breakfast/morning snack, lunch, and afternoon snack. Food diaries completed by parents will be used to assess children's dietary intake outside of child care. Parents will complete diary records on two weekdays (coinciding with the center visit) and one weekend day. The diary will prompt parents to record foods consumed, portion size, location, and time for each meal or snack. Follow-up phone calls will be conducted as needed to fill in any missing details. The combined DOCC and diary data will be analyzed with the Nutrition Data System for Research (NDSR) software in order to calculate children's daily intake of food groups, calories, and nutrients. Healthy Eating Index-2005 (HEI-2010) scores will be calculated for each child from these data.

Children's height and weight measurements will be collected by trained data collectors during the center site visit. This data (along with parent-reported child age and sex) will be used to calculate children's BMI, BMI percentile, and BMI z-score using standards and reference data provided by the Centers for Disease Control and Prevention (CDC 2010).

The food and physical activity environments of homes and child care centers will be assessed using the Home Self-administered Tool for Environmental assessment of Activity and Diet (HomeSTEAD) (Hales 2014) and the Environment and Policy Assessment and Observation (EPAO) (Ward 2008). HomeSTEAD is a self-administered survey that assesses characteristics of the home environment that influence children's diet and physical activity behaviors. The EPAO is an observation protocol that will provide similar data about the food and physical activity environments at child care centers. EPAO observations will be completed during the center visit by trained and certified data collectors. Data from HomeSTEAD and EPAO will be used to calculate scores for home and center nutrition and physical activity environments.

Parents and child care providers will also be asked to complete brief demographic surveys and health behavior screeners. Demographic surveys will assess standard characteristics like gender, age, race/ethnicity, marital status, household income, and employment. Center directors will also complete a demographic survey about the centers' current star rating, acceptance of child care subsidies, participation in the federally-funded Child and Adult Care Food Program (CACFP), and numbers, ages, and race/ethnicity of children enrolled. Given that the intervention targets parents' and child care providers' own health behaviors, the investigators will also collect self-reported data about provider and parent diet (fruit, vegetable, sweetened beverage intake), physical activity (frequency, and amounts of time spent in physical activities), and health status (weight and height), using several health behavior screeners.

Once all baseline measures are collected, centers will be randomly assigned (1:1) into the intervention or control arm. Centers in the intervention arm will immediately start implementation of Healthy Me, Healthy We. Centers in the control arm will receive the same intervention a year later (delayed).

Program Details/Intervention:

The program will be implemented center-wide (available to all 3-4 year old children and parents/families in each child care center in the intervention arm, regardless of participation in measurements). The campaign will begin in October and end in April of the same school year. At the start of the program center directors will notify parents about the program and hold a kick-off event. Following kick-off, the center will implement four units using materials provided by our research team. Each unit will last about six weeks, include a nutrition and physical activity theme, and incorporate visual cues, educational materials, and activities to deliver targeted messages.

Campaign components target both the child care center and home, two important spheres of influence that shape young children's diet and physical activity behaviors (Skouteris et al. 2011; Larsen et al. 2011). Engaging both spheres in a coordinated effort helps ensure that children receive consistent health messages. Messages will address the promotion and support of children's healthy diet and physical activity behaviors, while also encouraging child care staff and parents to adopt similar health behaviors. The messages within each unit will be informed by our conceptual model and address the following constructs: knowledge of current recommendations for children and adults, strategies for shaping the physical and social environment to promote good eating and physical activity habits, strategies for overcoming common barriers to healthy eating physical activity, and targets for making gradual behavior changes.

There are three key components to the program. First, is the commitment by the provider, the parent and the child, called the "Healthy We Promise." The provider, the parent and the child will each be asked to promise to take a "just try it" approach to healthy food and physical activity. Each family will receive a copy to sign and keep at home and each provider will be given a Healthy We Promise Poster to have children sign and display in their classroom.

The second component is classroom activities. A Unit Poster and Activity Cue Cards will be provided to facilitate these activities. The Unit Poster will be displayed in the classroom as a visual reminder to children about the overall goals of the current unit. Activity Cue Cards (about 12-16 cards) that match the Unit Poster will be given to providers. Each week, providers will select two cards and lead the classroom activities described.

The third component helps connect the classroom and home. A Healthy We Family Guide and Activity Tracker will go home with each child during the first week of each unit. The Family Guide has several components 1) introduction to the unit theme, 2) a Unit Guide tailored for at-home opportunities, 3) at-home versions of activities being completed in the classroom, 4) two to three recipes to try at home, and 5) expert tips about health and wellness. The Activity Tracker is designed to be placed on display at the child's home to allow for tracking of completed take-home activities. Throughout the unit, "Our Turn Tokens" are sent home whenever the provider completes an Activity Cue Card in the classroom. The Our Turn Token is intended to trigger parents to try the at-home version of the classroom activity.

At the end of the school year, each center will host a fun-festive gathering to celebrate all that providers, parents, and children have accomplished over the year. The event will include healthy food and fun, active games for the entire family.

Analysis:

Intervention impact on children's physical activity (i.e. minutes of non-sedentary physical activity) and diet quality (i.e. HEI score) will be assessed by comparing differences in mean changes from pre- to post-intervention between intervention and control arms using two-sided t-tests adjusted for clustering.

Our primary analyses will involve testing of each of these hypotheses under the intent-to-treat (ITT) principle (see section on missing data below) using Generalized Linear Mixed Models (GLMM) that will account for the correlation induced by the clustering of parents and children within childcare centers. Each GLMM (see below) will include a random intercept for childcare centers (b0) and fixed effects for the baseline value of the primary outcome (β1) and the intervention (β2) to test if the differences in mean changes in primary outcomes is zero, where β0 is the fixed intercept, and e is error.

Change in Primary Outcome9m = β 0 + β1 Primary Outcomebaseline + β2 Intervention + b0 + e

To further explore the effect of the intervention, the investigators will fit GLMMs that: 1) adjust for baseline covariates of interest, considered a priori, relevant to change in minutes of non-sedentary activity and HEI score; 2) adjust for baseline variables distributed differently between intervention groups; 3) test interaction terms between treatment group and other covariates; and 4) examine completers only.

Similar analyses will be used to examine change in child BMI, healthy weight attainment and maintenance, and change in scores on HomeSTEAD and EPAO. Demographic and health behavior data about the child care centers, providers, parents, and children will be analyzed descriptively, using frequencies, percentages, means, and standard deviations. In addition, the investigators will include this data as covariates in the GLMM models.

In alignment with RE-AIM (Reach Effectiveness Adoption Implementation Maintenance) (Glasgow et al. 1999), our process evaluation plan will include assessment of reach, effectiveness, adoption, implementation, and maintenance. These process measures will allow a fuller understanding of study results, how the program can be improved, and the potential for dissemination and sustainability.

ELIGIBILITY:
Inclusion Criteria:

Child Care Centers:

* Have 7-12 parent-child dyads willing to take part
* Have a Three, Four, or Five Star Rating OR GS110-106
* Serve lunch
* Have 3-4 year old classroom teachers that speak/write in English

Providers

* Teachers must teach in the 3-4 year old classrooms.
* Center directors and teachers must be able to read and speak English.

Parent-Child Dyad:

* Primary caregivers must have at least one 3-4 year old child enrolled in the participating center.
* Only one parent/primary caregiver will be eligible to participate.
* Can be male or female.
* Primary caregivers must be able to read and speak English.
* Special needs children must not have a chronic health issue that severely impacts their diet or physical activity.

Exclusion Criteria:

Child Care Centers:

* Serve special needs children exclusively
* Serve only non-English speaking families

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2293 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in child physical activity | Measures collected 3-10 weeks prior to start of intervention and 1-8 weeks post intervention
  Physical activity of 3-4 year old children will be assessed via accelerometry using ActiGraph monitors worn over the right hip for 7 days. Age-appropriate cut-points will be applied to calculate minutes of non-sedentary activity.
Change in child diet quality | Measures collected 3-10 weeks prior to start of intervention and 1-8 weeks post intervention
  Dietary intakes of 3-4 year old children will be assessed via direct observation of foods eaten at child care and parent report of foods eaten outside of child care. These dietary intake data will be used to calculate Healthy Eating Index scores as an indication of diet quality.

SECONDARY OUTCOMES:
Change in child weight | Measures collected 3-10 weeks prior to start of intervention and 1-8 weeks post intervention
  Height and weight of 3-4 year old children will be measured by trained staff. These data will be used to calculate children's body mass index (BMI). CDC growth charts and parent-report of child's sex and date of birth will then used to calculate BMI percentile, BMI z-score, and weight category (underweight, normal weight, overweight).
Change in nutrition and physical activity environments in homes and child care centers | Measures collected 3-10 weeks prior to start of intervention and 1-8 weeks post intervention
  The home environment will be assessed with HomeSTEAD, a self-administered survey completed by parents. The child care environments will be assessed with the Environment and Policy Assessment and Observation (EPAO), a measurement protocol conducted by trained data collectors during an onsite visit to the center.

CONTACTS AND LOCATIONS:
Overall Officials: Dianne S Ward, EdD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States